CLINICAL TRIAL: NCT01680458
Title: Special Investigation Of Fluconazole For Pediatric Subjects
Brief Title: Diflucan Research For Infant Evaluation Of Antifungal Treatment And Prophylaxis Medication
Acronym: DREAM
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A0561022
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Deep Mycosis
Keywords: antifungal treatment; prophylaxis; administration; Japanese; infants; fluconazole; Diflucan; Regulatory Post Marketing Commitment Plan.
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- fluconazole: Infant Subjects who are treated with fluconazole
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Fluconazole — Candidiasis infection: The recommended dosage in children is 3 mg/kg once daily.
  Cryptococcal infection: The recommended dosage in children is 6 mg/kg once daily. A dosage of 12 mg/kg once daily may be used, based on medical judgment of the patient's response to therapy.
  Prophylactic administration for deep mycosis on Hematopoietic stem cell transplantation: The recommended dosage in children is 12 mg/kg once daily.
  Absolute doses exceeding 600 mg/day are not recommended.
  Other Names: Diflucan

SUMMARY:
To collect the efficacy and safety information of fluconazole on infant subjects related to their appropriate use in daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female under age of seven patients who are prescribed fluconazole (Diflucan) for antifungal treatment or prophylaxis administration.

Exclusion Criteria:

* Subject of seven years or more who have been prescribed fluconazole.

Ages: 0 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The patients whom an investigator involving A0561022 prescribes the fluconazole (Diflucan).
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0561022&StudyName=Diflucan%20Research%20For%20Infant%20Evaluation%20Of%20Antifungal%20Treatment%20And%20Prophylaxis%20Medication

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluconazole: Pediatric participants aged less than 7 years at the start of administration received fluconazole according to Japanese package insert.
Period: Overall Study
Arm/Group | Fluconazole
Started | 30
Completed | 27
Not Completed | 3
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Population: In total, 30 participants were enrolled in the study. Of the 30 participants, a total of 3 participants were excluded from the baseline analysis because of protocol violation.
Arm/Group | Fluconazole
Number analyzed (Participants) | 27
Age, Customized [Number; unit: Participants]
  Less than 4 weeks | 1
  4 weeks to less than 1 year | 4
  1 to less than 7 years | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 9
Reason for administration, Treatment/Prophylaxis [Number; unit: Participants]
  Treatment | 2
  Prophylaxis | 25

OUTCOME MEASURES:

1. Secondary Outcome: Clinical Efficacy Rate
Description: Clinical effect of treatment was evaluated based on the clinical course excluding mycological effect as follows: (1) effective, (2) ineffective, or (3) unevaluable. Clinical efficacy rate was calculated as follows and presented along with the corresponding exact 2-sided 95% CI. Clinical efficacy rate (%) = (Number of responders in evaluation of clinical effect) / (Number of participants available for clinical efficacy evaluation) x 100.
Time Frame: MAX 13 Weeks
Population: Efficacy analysis set for treatment comprised of participants in safety analysis set (SAS) who had started to receive fluconazole for the treatment and had been evaluated for the clinical effect.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fluconazole
Number analyzed (Participants) | 2
Percentage of participants | 100 [2.50 to 100.00]

2. Secondary Outcome: Fungi Eradication Rate
Description: Mycological effect of treatment was evaluated as follows: (1) eradicated; the causative fungi detected from the lesion before treatment became undetectable, (2) presumably eradicated; the lesion was improved and sampling of causative fungi became impossible, (3) decreased; the causative fungi were decreased, (4) unchanged; no change was observed in the causative fungi, (5) increased; the causative fungi were increased (including microbial substitution), and (6) indeterminate; the clinical follow-up was inadequate, causative fungi were undetectable, or mycological test was not performed. Fungi eradication rate was calculated as follows. Fungi eradication rate (%) = (Number of participants evaluated as "eradicated" or "presumably eradicated") / (Number of participants available for mycological efficacy evaluation) x 100
Time Frame: MAX 13 Weeks
Population: Mycological analysis set for treatment comprised of participants in SAS with the final diagnosis of deep mycosis, who had started to receive fluconazole for the treatment and had been evaluated for the mycological effect.
Measure: Number; unit: Percentage of participants
Arm/Group | Fluconazole
Number analyzed (Participants) | 2
Percentage of participants | 0 [2.50 to 100.00]

3. Secondary Outcome: Onset Rate of Deep Mycosis
Description: Efficacy of deep mycosis prophylaxis was evaluated by the presence or absence of deep mycosis onset during the observation period. Onset rate of deep mycosis was calculated as follows and presented along with the corresponding exact 2-sided 95% CI. Onset rate of deep mycosis (%) = (Number of participants with deep mycosis onset by target fungi) / (Number of participants available for prophylactic efficacy evaluation) x 100.
Time Frame: MAX 13 Weeks
Population: Efficacy analysis set for prophylaxis comprised of participants in SAS who had started to receive fluconazole for the prophylaxis and had been evaluated for the presence or absence of deep mycosis onset.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fluconazole
Number analyzed (Participants) | 25
Percentage of participants | 0 [0.00 to 13.72]

4. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to fluconazole in a participant who received fluconazole. Relatedness to fluconazole was assessed by the investigator and sponsor (Pfizer Japan Inc.).
Time Frame: MAX 13 Weeks
Population: SAS comprised of participants who had met the inclusion criteria and had received fluconazole at least once.
Measure: Number; unit: Participants
Arm/Group | Fluconazole
Number analyzed (Participants) | 27
Participants | 1 [0.00 to 13.72]

5. Primary Outcome: Number of Participants With Treatment-Related Serious Adverse Events
Description: A treatment-related adverse event was any untoward medical occurrence attributed to fluconazole in a participant who received fluconazole. A treatment-related serious adverse event was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Relatedness to fluconazole was assessed by the investigator and sponsor (Pfizer Japan Inc.).
Time Frame: MAX 13 Weeks
Population: SAS comprised of participants who had met the inclusion criteria and had received fluconazole at least once.
Measure: Number; unit: Participants
Arm/Group | Fluconazole
Number analyzed (Participants) | 27
Participants | 0 [0.00 to 13.72]

6. Primary Outcome: Number of Participants With Treatment-Related Adverse Events Unexpected From Japanese Package Insert
Description: A treatment-related adverse event was any untoward medical occurrence attributed to fluconazole in a participant who received fluconazole. Expectedness of the adverse event was determined according to the Japanese package insert. Relatedness to fluconazole was assessed by the investigator and sponsor (Pfizer Japan Inc.).
Time Frame: MAX 13 Weeks
Population: SAS comprised of participants who had met the inclusion criteria and had received fluconazole at least once.
Measure: Number; unit: Participants
Arm/Group | Fluconazole
Number analyzed (Participants) | 27
Participants | 0 [0.00 to 13.72]

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Fluconazole
Serious Adverse Events (participants affected / at risk) | 2/27
Other Adverse Events (participants affected / at risk) | 9/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluconazole (N=27)
Skin infection (Infections and infestations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluconazole (N=27)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1)
Feeding disorder neonatal (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 2 (2)
Catheter site erythema (General disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Mucous membrane disorder (General disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.